CLINICAL TRIAL: NCT07279870
Title: RandomIsed sTudy of Physiologic cArdiac stimuLation in patIents With Atrio-ventricular Conduction Disease: the ITALIA Study
Brief Title: RandomIsed sTudy of Physiologic cArdiac stimuLation in patIents With Atrio-ventricular Conduction Disease
Acronym: ITALIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITALIA; 533/2025/Sper/AOUBo (Other: Comitato Etico AVEC)
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Atrioventricular Block
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conduction System Pacing (CSP) (Experimental): CSP occurs at the left endocardic surface of the interventricular septum hence specifically designed delivery catheters are used to advance the ventricular lead across the septum until its left-sided edge, where the Left Bundle is located.
  Interventions: Procedure: Conduction System Pacing (CSP)
- Conventional System Pacing/Right Ventricular (RV) Pacing (Active Comparator): RV pacing delivered either at the RV apex or RV septum. RV pacing is delivered by single chamber or dual chamber pacemakers depending on patients' rhythm (sinus or AT/AF) according to well-established clinical practice as described in the EHRA recommendtions
  Interventions: Procedure: Right Ventricular (RV) Pacing

INTERVENTIONS:
Procedure: Conduction System Pacing (CSP) — CSP occurs at the left endocardic surface of the interventricular septum hence specifically designed delivery catheters are used to advance the ventricular lead across the septum until its left-sided edge, where the Left Bundle is located. To determine whether CSP has been achieved, a standard 12-lead electrocardiogram (ECG) is continuously recorded.
  Arms: Conduction System Pacing (CSP)
Procedure: Right Ventricular (RV) Pacing — RV pacing delivered either at the RV apex or RV septum. RV pacing is delivered by single chamber or dual chamber pacemakers depending on patients' rhythm (sinus or AT/AF) according to well-established clinical practice as described in the EHRA recommendtions
  Arms: Conventional System Pacing/Right Ventricular (RV) Pacing

SUMMARY:
Study objective is to assess whether stimulation of the conduction system reduces cardiac decompensation events in patient follow-up, and how applicable this is in clinical practice and also to determine the impact of the studied interventions in terms of quality of life and cost-effectiveness for the treatment of patients with atrioventricular block. 1260 adult patients who are candidates for pacemaker implantation for the treatment of atrioventricular conduction disease will be randomised to stimulation of the conduction system or to the conventional stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with AV block in either sinus rhythm (SR) or permanent atrial tachycardia/atrial fibrillation (AT/AF), or with slow AV conduction during AT/AF, or undergoing AV node ablation + ventricular stimulation
* male and female
* acquired informed consent

Exclusion Criteria:

* Class I indication to Implantable Cardioverter Defibrillator (ICD) or to Cardiac Resynchronization Therapy (CRT)
* Ejection Fraction < 35%
* Life expectancy < 2 years
* Participation in another clinical trial which might impact on the study outcome
* Pregnancy, except as "In the event of an ongoing pregnancy, the doctor and patient will jointly assess, on a case-by-case basis and in the best interests of the patient, whether to propose participation in the study (random assignment to one of the two stimulation techniques) or to proceed as per clinical practice (assignment to one of the two stimulation techniques by the doctor). A screening log file of all eligible patients will be recorded, detailing the reason/s for non-randomization."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1260 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Heart failure | 36 months after the PM implant
  composite endponit of: number of HF events, HF hospitalizations and HF non-pharmacological interventions

SECONDARY OUTCOMES:
number of HF events | 36 months after the PM implant
  number of HF events
HF hospitalizations | 36 months after the PM implant
  HF hospitalizations
HF non-pharmacological interventions | 36 months after the PM implant
  HF non-pharmacological interventions

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Biffi, MD, Principal Investigator — IRCCS AOUBO Policlinico di Sant'Orsola
Locations (13):
- Italy (13):
  - Azienda Ospedal iera "Card. G. Panico", Bari
  - Azienda Ospedaliero-Universitaria Policlinico "G. Rodolico -San Marco", Catania
  - Azienda Ospedalie ro-Universitaria di Ferrara, Ferrara
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara, Novara
  - Azienda Sanitaria locali di Asti Ospedale Cardinal Massaia, Novara
  - Azienda Ospedaliero-Univeritaria di Palermo - Policlinico Giaccone, Palermo
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Azienda Ospedaliera Santa Maria della Misericordia, Perugia
  - Policlinico Casilino, Roma
  - Ospedale di Rovigo Aulss 5 Polesana, Rovigo
  - Città delle Salute e della Scienza di Torino. Dipartimento Cardiovascolare e Toracico, Torino
  - APSS Trento - Ospedale S. Maria del Carmine di Rovereto, Trento